CLINICAL TRIAL: NCT04794907
Title: Retinal Care Data Repository
Status: Not yet recruiting | Type: Observational
Sponsor: Retinal Care Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-PLN-003
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Retinopathy; Age Related Macular Degeneration
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DR: Patients with diabetes
  Interventions: Other: Observation
- AMD: Patients age 55 and older
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patient data will be collected from eye exams, surveys and medical record review.

SUMMARY:
The Retinal Care Data Repository's primary objective is to make data available for Retinal Care to develop algorithms that improve the care of people with retinal diseases.

DETAILED DESCRIPTION:
The initial focus is to develop algorithms that prevent, delay the progression, or improve treatment of diabetic retinopathy (DR) and age-related macular degeneration (AMD). Examples include but are not limited to: describing the incidence, prevalence, and severity distribution of DR and AMD in the overall population and subgroups; diagnosing specified severity thresholds for DR and AMD; predicting the development and progression of DR and AMD for the overall population, subgroups, and individuals; and recommending tests and treatments to prevent or delay the progression of DR and AMD for the overall population, subgroups, and individuals.

Data will be collected retrospectively and prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes or age 65 years and older

Exclusion Criteria:

* None

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The DR cohort includes any patient with diabetes. The AMD cohort includes patients 55 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Risk Stratification | Decade
  Predict the participant's risk of developing specific severity levels of DR and AMD

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Fransen, Principal Investigator — Retinal Care Inc.

IPD SHARING:
Plan to Share IPD: Undecided